CLINICAL TRIAL: NCT03371433
Title: Association Between Soft Drink Consumption and Osteoporotic Fractures Among Postmenopausal Women: The Women´s Health Initiative
Brief Title: Soft Drinks and Osteoporosis in WHI Participants
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Pedro Kremer, MD, MPH, Doctoral Student, University of California, San Diego
Other Study IDs: 170149XX
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Osteoporosis; Diet Habit
Keywords: Osteoporosis; Hip Fractures; Soft Drinks
MeSH Terms: conditions — Osteoporosis; Feeding Behavior; Hip Fractures | interventions — Carbonated Beverages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Soft drinks — Caffeine and Caffeine free soft drinks

SUMMARY:
Osteoporotic fractures, as a consequence of a reduced mineral bone density (BMD) represents a major public health problem. The lifetime risk of fractures exceeds 40% for women and 13% for men. At least ten different individual characteristics have already been proposed, evaluated, and some of them accepted as risk factors. Some of those risk factors were compiled in a tool developed by the World Health Organization in order to predict the ten-risk for a new fracture, even without considering BMD in that prediction . Increased consumption of carbonated soft drinks has been reported to have associations to a lower bone mineral density and an increment in bone fractures among young and also elder subjects.

However, some prospective studies have not found any significant associations and others suggested that risk is only increased for some kinds of beverages, like cola beverages, but not to the entire universe of soft drinks. In this sense, a large prospective analysis performed on 1413 women and 1125 men from the Framingham Offspring Cohort, analyzed- the relation between soft drinks consumption and BMD at the spine and 3 hip sites. Cola intake was associated with significantly lower BMD at each hip site, but not the spine, in women but not in men. Similar results were observed for diet cola and, although weaker, for decaffeinated cola. No significant relations between non-cola carbonated beverage consumption and BMD were observed.

In spite of the fact that reduced bone mineral density and osteoporotic fractures represent an increasing burden of disease and disability in postmenopausal women, most of the studies performed in this population used BMD as primary outcome, and not common osteoporotic fractures (e.g. hip, spine or wrist). Therefore, there is no conclusive evidence of a potential causal association between soft drinks (cola and non-cola) and fractures in a population in which osteoporotic fractures hold the highest incidence.

This research proposal is based on using the Women Health Initiative data to analyze the relation between cola and non-cola soft drinks consumption on common osteoporotic fractures. BMD will be considered a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* More than one day of follow up
* Dietary information on soft drinks

Exclusion Criteria:

Previous hip fracture

Ages: 50 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The WHI is an ongoing national study that enrolled 161,808 postmenopausal women aged 50-79 at baseline, enrolled during 1993-1998. Data collection at screening and enrollment included questionnaires completed by self-report or interview, physical examination, and blood specimen collection. Information on soda intake (total, caffeinated and caffeine-free) was collected at the sixth follow-up year in the OS among 79,885 women who form the baseline study population for this analysis. After exclusion of participants who had incomplete exposure information (n=5,413), had previous history of hip fracture (n=471), or less than one day of follow up after Year 6 (n=1659), a cohort of 72,342 participants contributing 700,388 person/years of follow-up was used for the prospective analysis. All participants provided informed consent at baseline and subsequently for extended follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 79885 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Lumbar spine osteoporosis | median 16 years
  Bone mineral density lumbar spine measured in grams/square centimeters
Total hip osteoporosis | median 16 years
  Bone mineral density at the total hip measured in grams/square centimeters
Hip fractures | median 16 years
  Number of participants that suffered a hip fracture

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnell O, Kanis JA. An estimate of the worldwide prevalence, mortality and disability associated with hip fracture. Osteoporos Int. 2004 Nov;15(11):897-902. doi: 10.1007/s00198-004-1627-0. Epub 2004 May 4. PMID 15490120
- [Background] Park S, Xu F, Town M, Blanck HM. Prevalence of Sugar-Sweetened Beverage Intake Among Adults--23 States and the District of Columbia, 2013. MMWR Morb Mortal Wkly Rep. 2016 Feb 26;65(7):169-74. doi: 10.15585/mmwr.mm6507a1. PMID 26914018
- [Background] Kim SH, Morton DJ, Barrett-Connor EL. Carbonated beverage consumption and bone mineral density among older women: the Rancho Bernardo Study. Am J Public Health. 1997 Feb;87(2):276-9. doi: 10.2105/ajph.87.2.276. PMID 9103110
- [Background] Ogur R, Uysal B, Ogur T, Yaman H, Oztas E, Ozdemir A, Hasde M. Evaluation of the effect of cola drinks on bone mineral density and associated factors. Basic Clin Pharmacol Toxicol. 2007 May;100(5):334-8. doi: 10.1111/j.1742-7843.2007.00053.x. PMID 17448120
- [Background] Tucker KL, Morita K, Qiao N, Hannan MT, Cupples LA, Kiel DP. Colas, but not other carbonated beverages, are associated with low bone mineral density in older women: The Framingham Osteoporosis Study. Am J Clin Nutr. 2006 Oct;84(4):936-42. doi: 10.1093/ajcn/84.4.936. PMID 17023723
- [Background] Fung TT, Arasaratnam MH, Grodstein F, Katz JN, Rosner B, Willett WC, Feskanich D. Soda consumption and risk of hip fractures in postmenopausal women in the Nurses' Health Study. Am J Clin Nutr. 2014 Sep;100(3):953-8. doi: 10.3945/ajcn.114.083352. Epub 2014 Aug 6. PMID 25099544
- [Background] Chen Z, Kooperberg C, Pettinger MB, Bassford T, Cauley JA, LaCroix AZ, Lewis CE, Kipersztok S, Borne C, Jackson RD. Validity of self-report for fractures among a multiethnic cohort of postmenopausal women: results from the Women's Health Initiative observational study and clinical trials. Menopause. 2004 May-Jun;11(3):264-74. doi: 10.1097/01.gme.0000094210.15096.fd. PMID 15167305
- [Background] Fitzpatrick L, Heaney RP. Got soda? J Bone Miner Res. 2003 Sep;18(9):1570-2. doi: 10.1359/jbmr.2003.18.9.1570. No abstract available. PMID 12968665
- [Background] Cuomo R, Sarnelli G, Savarese MF, Buyckx M. Carbonated beverages and gastrointestinal system: between myth and reality. Nutr Metab Cardiovasc Dis. 2009 Dec;19(10):683-9. doi: 10.1016/j.numecd.2009.03.020. Epub 2009 Jun 6. PMID 19502016
- [Background] Design of the Women's Health Initiative clinical trial and observational study. The Women's Health Initiative Study Group. Control Clin Trials. 1998 Feb;19(1):61-109. doi: 10.1016/s0197-2456(97)00078-0. PMID 9492970
- [Background] Wyshak G, Frisch RE. Carbonated beverages, dietary calcium, the dietary calcium/phosphorus ratio, and bone fractures in girls and boys. J Adolesc Health. 1994 May;15(3):210-5. doi: 10.1016/1054-139x(94)90506-1. PMID 8075091